CLINICAL TRIAL: NCT04257175
Title: Giving CAR-T CD19 Transgenic T Cells for Acute Myeloid Leukemia Patients (AML) With t 8:21 and CD19 Expression
Brief Title: CAR-T CD19 for Acute Myelogenous Leukemia With t 8:21 and CD19 Expression
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof Arnon Nagler, M.D., M.Sc, Professor of Medicine Tel Aviv University, Director Hematology Division, Chaim Sheba Medical Center, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6482-19-SMC
Record Dates: First submitted 2020-01-20; First posted 2020-02-05 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Chimeric antigen receptors; Mixed phenotype acute leukemia; T cells.
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyclophosphamide, Flodarabine,CAR-T cells (Experimental): The appropriate participants will undergo lymhopheresis to collect lymphocytes from PBMC peripheral blood. CAR T CD19 cells will be produced. The participants will receive cyclophosphamide 300 mg / m² and flodarabine 30 mg / m² lymphodeplition intravenously daily for 3 days.
  The CAR-T CD19 cells will be given on the 5 to 7 day post lymphodeplition .
  Interventions: Biological: CAR-T CD19

INTERVENTIONS:
Biological: CAR-T CD19 — The CAR-T infusion will be given in IV infusion. The target dose is 1 X 106 positive CAR / kg T cells (range: 0.5-1.5X 106 CAR / kg positive T cells).

SUMMARY:
Chimeric antigen receptor (CAR-T) engineered T cells against the CD19 protein have been shown to be effective against acute lymphoma and lymphocytic leukemia and are approved by the US (FDA), European (EMA) and Health Basel.

However, little information exists on using CD19CAR for treatment of recurrent or irresponsible to previous treatment acute myeloid leukemia.

The proposed study will include patients with recurrent disease or those with disease irresponsible to common treatments and they will be treated with CAR-T CD19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent acute myeloid leukemia (AML) including those after bone marrow transplantation or not responding to previous therapy, who have exhausted other approved relevant therapies such as chemotherapy protocols that are ineffective and with high toxicity, or FLT3 inhibitors in patients with FLT3 .

Exclusion Criteria:

* Heart disease including severe heart failure (NYHA III-IV), recent MI or CABG surgery (in previous six months), severe ventricular rhythm abnormalities, non ischemic heart disease, LVEF less than 45%
* Active involvement of CNS
* Active infection
* Pregnancy or lactation
* Graft versus host disease III-IV grade - Stroke or seizure in the last six months before treatment
* A positive result for the HIV infection (serum)
* Active hepatitis infection
* Life-threatening allergies to cyclophosphamide or fludarabine
* No informed consent signed by candidate
* Candidate enrolled in other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The change in the peripheral blood counts and differential | Within two years from the introduction of the CAR-T CD19
  Will be evaluated by Coulter counter
The change in the antigen expression on the leukemic blasts | Within two years from the introduction of the CAR-T CD19
  Will be evaluated by FACS
The change in the measurable residual disease | Within two years from the introduction of the CAR-T CD19
  Will be evaluated by PCR
The change in the chromosomal translocations and aberrations | Within two years from the introduction of the CAR-T CD19
  Will be evaluated by cytogenetics and FISH

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel